CLINICAL TRIAL: NCT03381508
Title: Retrospective Analysis of the Determinants of Air Leakage in a Population of Obstructive Sleep Apnea Syndrome Treated With Continuous Positive Airway Pressure
Brief Title: Air Leakage Under Continuous Positive Airway Pressure
Acronym: SAS-leak-1
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0429
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: CPAP; masks; unintentional leak; leakage
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: The study population corresponds to patients with obstructive sleep apnea syndrome treated via continuous positive pressure and monitored according to usual practice with the latest Brizzy device.
  Intervention: Brizzy continuous positive pressure device
  Interventions: Device: Brizzy continuous positive pressure device

INTERVENTIONS:
Device: Brizzy continuous positive pressure device — Patients are treated with the Brizzy continuous positive pressure device, including pneumotachograph.

SUMMARY:
The software embedded in recent continuous positive pressure devices enables the analysis of the level of leakage that occurs during treatment around the mask or from the mouth. However, there is no clear threshold defining when it would be appropriate to implement means for correcting these leaks. In addition, the calculation methods used to detect/measure leaks and the terminology used vary according to the manufacturers of continuous pressure devices, which also complicates the clinical interpretation of the leakage reports provided by the various devices.

In daily practice, when a patient complains of unintentional leakage, technicians adjust the mask, replace the nasal-mask by an oro-nasal mask or install a chinstrap. Nevertheless, those strategies are not always effective in reducing leakage or patient's complaints. A better understanding of the mechanisms beyond leak appearance for a given patient could lead to individualised leak-treatment solutions. Pressure level, mandibular behaviour, respiratory effort, sleep position or sleep stages may contribute to leak emergence.

A recent exploratory study has proposed a genuine analysis method of determining factors of unintentional-leaks using polysomnographic recordings in OSA patients treated with automatic Continuous Positive Airway Pressure (auto-CPAP). Based on the same methodology, the NOMICS company (Liège, Belgium) has developed a polygraphic device (Brizzy®) recording unintentional leakage during auto-CPAP treatment and providing an etiological analysis of unintentional-leaks via a software named APIOS.

Due to the innovative nature of the analysis, it appears necessary to validate it onto a population of OSA patients treated with auto-CPAP. Also, to our knowledge, there is no descriptive data of the distribution of the determinants of unintentional leaks in such a population. From this perspective, the investigators aim to retrospectively analyse some polygraphic recordings that have been performed with the Brizzy® on OSA patients treated with auto-CPAP.

The primary objective of this study is to identify and describe the determinants of unintentional leaks for a population of patients with OSA and treated with an auto-CPAP device

DETAILED DESCRIPTION:
The secondary objectives are:

1. to evaluate the concordance of the determinants of leaks according to different leak thresholds (0 l/min ; 5l/min ; 10l/min : 20l/min).
2. to describe any technical problems that arise in relation to the analysis of leaks in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Sleep recordings from patients with OSA treated via auto-CPAP and monitored with Brizzy® device (including measures of non-intentional leaks) between June 1st and December 31th, 2017.

Exclusion Criteria:

* The patient opposes the usage of his/her data
* Minors or adults under any kind of guardianship
* Fixed pressure
* Bilevel positive airway pressure devices
* Adaptive servo-ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to patients (all meeting eligibility criteria) with obstructive sleep apnea syndrome treated via continuous positive pressure and monitored according to usual practice with the latest Brizzy device.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Mouth-opening odds ratio | day 0 (transversal study)
  For each patient presenting with an unintentional leak, determination of odds ratios for mouth-opening.
Auto-CPAP pressure level odds ratio | day 0 (transversal study)
  For each patient presenting with an unintentional leak, determination of odds ratios for Auto-CPAP pressure level
Sleep position odds ratio | day 0 (transversal study)
  For each patient presenting with an unintentional leak, determination of odds ratios for sleep position
Respiratory effort (increase in the Jawac signal > 0.3 mm) odds ratio | day 0 (transversal study)
  For each patient presenting with an unintentional leak, determination of odds ratios respiratory effort

SECONDARY OUTCOMES:
Epworth scale score | day 0 (transversal study)
Pichot scale | day 0 (transversal study)
Occurrence of nasal obstruction | day 0 (transversal study)
Occurrence of mouth dryness | day 0 (transversal study)
Occurrence of nasal dryness | day 0 (transversal study)

OTHER OUTCOMES:
Type/brand of mask and device used | day 0 (transversal study)
Presence of heated humidifier | day 0 (transversal study)
Presence of chinstraps. | day 0 (transversal study)
The Brizzy output | day 0 (transversal study)
Mask pressure as measured by Brizzy | day 0 (transversal study)
Presence/absence of technical problems that arise in relation to the analysis of leaks | day 0 (transversal study)
Presence/absence of a comorbidity | day 0 (transversal study)
Presence of a psychotropic treatment | day 0 (transversal study)
Presence of a treatment of nasal problem | day 0 (transversal study)
Anterior ORL surgery | day 0 (transversal study)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christian Borel, PhD, Principal Investigator — University Hospital, Grenoble; Nicolas Molinari, PhD, Study Director — University Hospital, Montpellier
Locations (3):
- France (3):
  - Polyclinic Saint-Privat, Boujan-sur-Libron
  - University Hospital of Grenoble, Grenoble
  - Hôpital Arnaud de Villeneuve, Montpellier

REFERENCES:
- [Result] Lebret M, Arnol N, Martinot JB, Lambert L, Tamisier R, Pepin JL, Borel JC. Determinants of Unintentional Leaks During CPAP Treatment in OSA. Chest. 2018 Apr;153(4):834-842. doi: 10.1016/j.chest.2017.08.017. Epub 2017 Aug 26. PMID 28847549
- [Result] Lebret M, Jaffuel D, Suehs CM, Mallet JP, Lambert L, Rotty MC, Pepin JL, Matzner-Lober E, Molinari N, Borel JC. Feasibility of Type 3 Polygraphy for Evaluating Leak Determinants in CPAP-Treated OSA Patients: A Step Toward Personalized Leak Management. Chest. 2020 Nov;158(5):2165-2171. doi: 10.1016/j.chest.2020.05.593. Epub 2020 Jun 13. PMID 32544491